CLINICAL TRIAL: NCT03030534
Title: Research Protocol On Developing an Integrated Technology-Moderated Institutional Health Promotion Model (ITIHPM)for Use in Nigeria Universities
Brief Title: Research Protocol On Developing an Integrated Technology-Moderated Institutional Health Promotion Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Responsible Party: Principal Investigator, Elizabeth M. Joseph-Shehu, Principal investigator, University of KwaZulu
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DITIHPM-001
Record Dates: First submitted 2017-01-19; First posted 2017-01-25 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups. that is two locations (study centres) will be selected for the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Educational Package and software package
  Interventions: Combination Product: Educational package and software package
- Control group (Active Comparator): Health promotion tips
  Interventions: Other: Health promotion tips

INTERVENTIONS:
Combination Product: Educational package and software package — Using Information and communication technology to deliver health promoting activities
  Other Names: Health promotion lifestyle activities
  Arms: Experimental Group
Other: Health promotion tips — Give general information on health promotion
  Arms: Control group

SUMMARY:
The purpose of this study is to adopt an operational research approach that seeks to design, develop and pilot-test the health-promotion lifestyle model that will enhance health-promoting behaviour and lifestyle modification of university staff in Nigeria. The following are the hypotheses of the study:

1. There will be a significant difference in the pre and post intervention practices of health promoting lifestyle behaviours (behaviour specific cognition and affect) of NOUN staff
2. There will be significant association between the health promoting lifestyle behaviours (behavioural outcome) and health status of NOUN staff
3. There will be a significant difference in the pre-and post-intervention health promoting lifestyle behaviours (behavioural outcome) of staff of NOUN
4. There will be a significant difference in the pre-and post-intervention health status measure (specific health measurement indicators) of staff of NOUN

DETAILED DESCRIPTION:
Health promotion is advocated worldwide as being an efficient strategy to enhance quality of life and control the increasing prevalence of non-communicable diseases. health promoting lifestyle has been linked to high prevalence of most non-communicable diseases. Efficient and effective health promoting lifestyle practices is beneficial in prevention and control of non-communicable diseases, as well as improving the quality of life. World Health Organization has established workplace and schools as priority settings for health promotion in the 21st century as locus of reaching large number of audience. Workplace and schools also offer an ideal settings and infrastructure to support the health promoting activities that will improve the quality of life of workers and students. Information and communication technologies (ICTs) has made the world a global village, both young and old engages in one form of ICTs or the other. This study aims to adopt operational research approach to design, develop and pilot-test Integrated Technology-Moderated Institutional Health Promotion Model (ITIHPM) that will enhance health promoting behaviour and lifestyle modification of staff in Nigeria universities.

The objectives of the study are:

1. To determine the health-promoting behaviour of NOUN staff;
2. To assess the health status of NOUN staff;
3. To examine factors that influence the health promoting lifestyle behaviour of NOUN staff;
4. To assess institutional policies available to encourage NOUN staff to practise health -promoting lifestyles;
5. To assess resources available in the institution that encourage health-promoting behavior;
6. To examine protocols in place to ensure adoption of health-promoting behaviour and healthy lifestyle of NOUN staff;
7. To determine technology-moderated applications/platforms that would be useful in promoting knowledge and skills acquisition for health-promoting behaviour and lifestyle modifications among NOUN staff; and
8. To determine the impact of a technologically-based institutional health promotion model among NOUN staff.

Who can participate? All staff that are on the university pay roll in the selected study centres, irrespective of their age.

What does the study involve? Two study centres will be randomly selected from the six study centers selected during the first phase of the study. The two centres are randomly allocated into two groups two (experimental group and control group). The control group will receive tips on health promoting lifestyle practices, answer health promoting lifestyle profile questionnaire before giving the tips, have their weight, height, blood pressure, fasting blood sugar, abdominal circumference and hip circumference checked. The group will further answer the questionnaire and have their weight, height, blood pressure, fasting blood sugar, abdominal circumference and hip circumference checked at 6 weeks and at 12 weeks. While the experimental group will have four weeks training (educational package) on nutrition, exercise/physical activity, stress management, health responsibility, self-actualization and interpersonal relationship through seminar and symposium for 45-60 minutes 4 times in a week for the 4 weeks. At the beginning of the training database of all the participants will be created. This will include socio-demographic data and baseline health assessment that is related to the study (weight, height, blood pressure, fasting blood sugar, abdominal circumference and hip circumference). Participants will also answer questionnaire on health promoting lifestyle practice at the beginning of the training. The same procedure will be taken at week zero (immediately after the training), at 6 weeks and at 12 weeks. In the last two sections of the meeting, participants will be informed and intimate on the use of the software package and encourage them to ask questions. The participants will receive audio and video messages on health promoting lifestyle practices once in a week. The software application will be designed in a way that both the principal investigator and participants can interact at any time. The Technology-Moderated Institutional Health Promotion Model will also give opportunity to university staff to have assessed to a Community Health Nurse Specialist (health promotion expert) at every needed time. Four sessions of Focus Group Discussions among cohorts of staff will be conducted to identify barriers to healthy lifestyle practices using the developed model.

Primary outcome measures

1. Health promoting lifestyle practices of staff will be measured using health promoting lifestyle profile II at the beginning of the study.
2. Effective and efficient Health promoting lifestyle practices of staff will be measured using health promoting lifestyle profile II and mobile software application at zero week, 6 weeks and 12 weeks
3. Health status of staff will be measured using the following indicators: weight, height, blood pressure, fasting blood sugar, abdominal circumference and hip circumference at the beginning of the study, at zero week, 6 weeks and 12 weeks
4. Resources available in the university that will enhance health promoting lifestyle practices will be measured using interview guide and checklists at the beginning of the study Secondary outcome measures

1. Participants compliance to the intervention will be measured at 6 weeks and 12 weeks 2. Participants satisfaction with the intervention will be measured at 6 weeks and 12 weeks 3. Retention rate will be measured at 6 weeks and 12 weeks

The target number of participants in the pilot-testing phase is 185 Exclusion criteria

What are the possible benefits and risks of participating? We hope that the study will afford the participants the benefits of practicing health promoting lifestyle effectively and thereby help him/her to prevent non-communicable diseases (NCDs). In case the participant has been diagnosed with any NCDs, participating in this study will provide the individual with relevant information that will make him/her live a quality life. During the study if the health assessment reveals any deviation from normal, the individual will be referred to the school sickbay for appropriate treatment and the principal researcher will still follow the him/her up. The only risk anticipated in this study is that its demands the participants to be meticulous in adhering to all the health promotion activities, which are beneficial on the long to the participants.

ELIGIBILITY:
Inclusion Criteria:

* All staff of the university in the selected study centres
* Own a smartphone that can take the software application (experimental group)

Exclusion Criteria:

* Unwilling to participate in the study
* unable to use smartphone

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Changes in Health promoting lifestyle practices | Baseline, 6 weeks and 12 weeks
  health promoting lifestyle profile questionnaire consist of six subclass (Nutrition, Physical activity, Health responsibility, Stress management, interpersonal relationship, self-actualization) of health promoting lifestyle activities and self-designed mobile software application

SECONDARY OUTCOMES:
BMI in kg/m^2 | Baseline, at 6 weeks and 12 weeks
  Assess changes in BMI
Random blood glucose in mg/dl | Baseline, 6 weeks and 12 weeks
  Assess changes in participants blood glucose
Waist to Hip ratio (WHR) in cm | Baseline, 6 weeks and 12 weeks
  Assess changes in Waist to Hip ratio
Blood pressure in mmHg | Baseline, 6 weeks and 12 weeks
  Assess changes in participants blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Joseph-Shehu, MSc, Principal Investigator — University of KwaZulu-Natal, Durban, South Africa
Locations (1):
- National Open University of Nigeria, Abuja, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided
All data that will be beneficial to other researchers will be sheared through journal publication and workshops. No identifying data will be published.

REFERENCES:
- [Result] Şenol V, Ünalan D, Soyuer F, Argün M: The relationship between health promoting behaviors and quality of life in nursing home residents in Kayseri. Journal of Geriatrics 2014
- [Result] Chronic diseases and health promotion: Global Status Report on NCDs
- [Result] Oinas-Kukkonen H: Behavior change support systems: A research model and agenda. In: Persuasive Technology. edn.: Springer; 2010: 4-14.
- [Result] Cowdery J, Kindred J, Michalakis A, Suggs LS: Promoting health in a virtual world: Impressions of health communication messages delivered in Second Life. First Monday 2011, 16(9).
- [Result] Bock BC, Graham AL, Whiteley JA, Stoddard JL. A review of web-assisted tobacco interventions (WATIs). J Med Internet Res. 2008 Nov 6;10(5):e39. doi: 10.2196/jmir.989. PMID 19000979
- [Result] Koniak-Griffin D, Brecht ML, Takayanagi S, Villegas J, Melendrez M, Balcazar H. A community health worker-led lifestyle behavior intervention for Latina (Hispanic) women: feasibility and outcomes of a randomized controlled trial. Int J Nurs Stud. 2015 Jan;52(1):75-87. doi: 10.1016/j.ijnurstu.2014.09.005. Epub 2014 Sep 22. PMID 25307195
- [Result] Wikstrom K, Lindstrom J, Tuomilehto J, Saaristo TE, Helakorpi S, Korpi-Hyovalti E, Oksa H, Vanhala M, Keinanen-Kiukaanniemi S, Uusitupa M, Peltonen M. National diabetes prevention program (DEHKO): awareness and self-reported lifestyle changes in Finnish middle-aged population. Public Health. 2015 Mar;129(3):210-7. doi: 10.1016/j.puhe.2014.12.019. Epub 2015 Feb 26. PMID 25726122